CLINICAL TRIAL: NCT01438606
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of VSV-Indiana HIV Gag Vaccine Given Intramuscularly in Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Evaluating the Safety of and Immune Response to the VSV-Indiana HIV Vaccine in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 090; 11669 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- 1 x 10^4 PFU VSV-Indiana HIV gag vaccine (Group 1) (Experimental): Participants will receive 1 x 10^4 PFU of the study vaccine by intramuscular (IM) injection in each deltoid at baseline and Week 8. (1 x 10^4 PFU is the nominal dose; the actual dose is 4.6 x 10^3 PFU given as 2.3 x 10^3 PFU in each deltoid)
  Interventions: Biological: VSV-Indiana HIV gag vaccine
- Placebo injection (normal saline) (Group 1) (Placebo Comparator): Participants will receive placebo by IM injection in each deltoid at baseline and Week 8.
  Interventions: Biological: Placebo injection (normal saline)
- 1 x 10^5 PFU VSV-Indiana HIV gag vaccine (Group 2) (Experimental): Participants will receive 1 x 10^5 PFU of the study vaccine by IM injection in each deltoid at baseline and Week 8. (1 x 10^5 PFU is the nominal dose; the actual dose is 4.6 x 10^4 PFU given as 2.3 x 10^4 PFU in each deltoid)
  Interventions: Biological: VSV-Indiana HIV gag vaccine
- Placebo injection (normal saline) (Group 2) (Placebo Comparator): Participants will receive placebo by IM injection in each deltoid at baseline and Week 8.
  Interventions: Biological: Placebo injection (normal saline)
- 1 x 10^6 PFU VSV-Indiana HIV gag vaccine (Group 3) (Experimental): Participants will receive 1 x 10^6 PFU of the study vaccine by IM injection in each deltoid at baseline and Week 8. (1 x 10^6 PFU is the nominal dose; the actual dose is 4.8 x 10^5 PFU given as 2.4 x 10^5 PFU in each deltoid)
  Interventions: Biological: VSV-Indiana HIV gag vaccine
- Placebo injection (normal saline) (Group 3) (Placebo Comparator): Participants will receive placebo by IM injection in each deltoid at baseline and Week 8.
  Interventions: Biological: Placebo injection (normal saline)
- 1 x 10^7 PFU VSV-Indiana HIV gag vaccine (Group 4) (Experimental): Participants will receive 1 x 10^7 PFU of the study vaccine by IM injection in each deltoid at baseline and Week 8. (1 x 10^7 PFU is the nominal dose; the actual dose is 4.2 x 10^6 PFU given as 2.1 x 10^6 PFU in each deltoid)
  Interventions: Biological: VSV-Indiana HIV gag vaccine
- Placebo injection (normal saline) (Group 4) (Placebo Comparator): Participants will receive placebo by IM injection in each deltoid at baseline and Week 8.
  Interventions: Biological: Placebo injection (normal saline)
- 1 x 10^8 PFU VSV-Indiana HIV gag vaccine (Group 5) (Experimental): Participants will receive 1 x 10^8 PFU of the study vaccine by IM injection in each deltoid at baseline and Week 8. (1 x 10^8 PFU is the nominal dose; the actual dose is 3.4 x 10^7 PFU given as 1.7 x 10^7 PFU in each deltoid)
  Interventions: Biological: VSV-Indiana HIV gag vaccine
- Placebo injection (normal saline) (Group 5) (Placebo Comparator): Participants will receive placebo by IM injection in each deltoid at baseline and Week 8.
  Interventions: Biological: Placebo injection (normal saline)

INTERVENTIONS:
Biological: VSV-Indiana HIV gag vaccine — Administered IM in both deltoids at baseline and Week 8. Dose will vary depending on which group the participant is enrolled in.
  Arms: 1 x 10^4 PFU VSV-Indiana HIV gag vaccine (Group 1); 1 x 10^5 PFU VSV-Indiana HIV gag vaccine (Group 2); 1 x 10^6 PFU VSV-Indiana HIV gag vaccine (Group 3); 1 x 10^7 PFU VSV-Indiana HIV gag vaccine (Group 4); 1 x 10^8 PFU VSV-Indiana HIV gag vaccine (Group 5)
Biological: Placebo injection (normal saline) — Administered IM in both deltoids at baseline and Week 8.
  Arms: Placebo injection (normal saline) (Group 1); Placebo injection (normal saline) (Group 2); Placebo injection (normal saline) (Group 3); Placebo injection (normal saline) (Group 4); Placebo injection (normal saline) (Group 5)

SUMMARY:
The purpose of this study is to evaluate the safety and immune response to an HIV vaccine in HIV-uninfected adults. Study researchers will also determine the maximum dose of the vaccine that participants can safely receive.

DETAILED DESCRIPTION:
Many HIV vaccines that are in development use a virus vector to deliver the vaccine into the body's cells in order to elicit an immune response. Vesicular stomatitis virus (VSV) is a vector that has been studied in animals. As an HIV vaccine vector, it has been shown to prevent disease progression in monkeys infected with simian/human immunodeficiency virus (SHIV). This study will evaluate the safety and immune response to the VSV-Indiana (one type of VSV vector) HIV gag vaccine in healthy, HIV-uninfected adults. In addition, study researchers will determine the maximum dose of the vaccine that can be safely tolerated.

This study will enroll healthy, HIV-uninfected adults. Five groups of participants will be enrolled, with each subsequent group receiving a slightly higher dose of the vaccine. Within each group, participants will be randomly assigned to receive the study vaccine or a placebo vaccine. Study researchers will examine safety data and how participants react to the study vaccine before enrolling the next group of participants. At baseline and Week 8, participants will receive two injections of the study vaccine or placebo vaccine-one in each upper arm at each time point. At the baseline study visit, all participants will undergo a physical examination; mouth examination; a medical and medication history review; and saliva, blood, and urine collection. Female participants will also take a pregnancy test. Participants will complete questionnaires to assess mental status and receive counseling on HIV risk reduction and pregnancy prevention. After receiving the vaccine, participants will remain in the clinic for at least 30 minutes for observation and monitoring of side effects. For 7 days after the vaccination, participants will record any side effects in a symptom log.

Participants will attend study visits 3 days and 1 and 2 weeks after the baseline study visit, at Week 8 for the second vaccination, 3 days and 1 and 2 weeks after the Week 8 visit, and at Months 5 and 8. Follow-up study visits will include select baseline study procedures. Participants will be contacted annually for 3 years for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HVTN Clinical Research Site (CRS) and willing to be followed for the planned duration of the study
* Able and willing to provide informed consent
* Demonstrate understanding of this study by completing a questionnaire prior to first vaccination, with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required study visit
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required study clinic visit (excludes annual contacts for safety surveillance)
* In good general health as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as being at "low risk" of HIV infection
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female, greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell (WBC) count of 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets between 125,000 and 550,000/mm^3
* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and creatinine values less than or equal to institutional upper limits of normal
* Negative HIV-1 and -2 blood test: participants in the United States must have a negative Food and Drug Administration (FDA)-approved immunoassay (IA)
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV) or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine: negative urine glucose, negative or trace urine protein, and negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis must be within institutional normal range)
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Participants who were born female must agree to consistently use effective contraception from 21 days prior to study entry through the last required study clinic visit for sexual activity that could lead to pregnancy, or not be of reproductive potential, or be sexually abstinent. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required study clinic visit

Exclusion Criteria:

* Excessive daily alcohol use, frequent binge drinking, chronic marijuana abuse, or any other use of illicit drugs within the 6 months prior to study entry
* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B within the 12 months prior to study entry
* Untreated or incompletely treated syphilis infection
* HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 090 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the 5 years prior to study entry in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For potential participants who have received control/placebo in an experimental vaccine trial, the HVTN 090 PSRT will determine eligibility on a case-by-case basis. For potential participants who have received an experimental vaccine(s) greater than 5 years prior to study entry, eligibility for enrollment will be determined by the PSRT on a case-by-case basis.
* Immunosuppressive medications received within 168 days before first vaccination (Not excluded: [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or fewer with completion at least 30 days prior to study entry].)
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 12 months before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 090 study
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to study adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the 12 months prior to study entry
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* Hypertension:

  1. If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at study entry.
  2. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at study entry or diastolic blood pressure greater than or equal to 100 mm Hg at study entry.
* Body mass index (BMI) greater than or equal to 40 or BMI greater than or equal to 35 with two or more of the following criteria: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, known hyperlipidemia
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Cancer (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
* Seizure disorder (any history of seizure)
* Neurological or neuropsychiatric disorder that may interfere with the assessment of safety such as: frequent recurring headaches (e.g., a pattern of more than one headache per month affecting activities of daily living [ADLs]/work, frequent or severe/complicated migraines, cluster headaches), a chronic pain syndrome, dizziness, history of meningitis or encephalitis, cranial/spinal/peripheral neuropathy, limb weakness or paralysis, movement disorder, narcolepsy, stroke with sequelae, moderate/severe major depressive disorder, or moderate/severe bipolar disorder
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the study. Specifically excluded are people with psychoses within the 3 years prior to study entry, ongoing risk of suicide, or history of suicide attempt or gesture within the 3 years prior to study entry.
* Pregnant or breastfeeding
* Lives with or cares for any of the following: a person less than or equal to 2 years of age or greater than 65 years of age, a person who is immunocompromised (at risk of opportunistic infection), or a person with a chronic lung disease (such as cystic fibrosis or requiring daily oral corticosteroids or home oxygen)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in frequency and severity of local injection site reactogenicity signs and symptoms | Measured at Days 0, 1, 2, 4, 5, 6, 7, 60, 61, 62, 63, 64, 65, 66, and 67
  Pain, tenderness, erythema, induration, and maximum severity of pain and/or tenderness; frequency and severity of systemic reactogenicity signs and symptoms: fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and maximum severity of systemic symptoms
Frequency of adverse events (AEs) categorized by Medical Dictionary for Regulatory Activities (MedDRA) body system | Participants will be followed for the duration of the study, an expected average of 8 months
  Frequency of AEs categorized by MedDRA body system, MedDRA preferred term, severity and assessed relationship to study products; detailed description of all serious adverse events (SAEs)
Change in distribution of values of safety laboratory measures | Measured at Days 3, 5, 9, and 140
  White blood cells (WBCs), neutrophils, lymphocytes, hemoglobin, alkaline phosphatase, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatinine at baseline and at follow-up visits postvaccination
Number of participants with early discontinuation | Participants will be followed for the duration of the study, an expected average of 8 months
  Number of participants with early discontinuation of vaccinations and reason for discontinuation

SECONDARY OUTCOMES:
Change in response rates of CD4 T-cell responses | Measured at Days 7, 14, 68, and 70
  Response rates of CD4 T-cell responses measured by intracellular cytokine staining (ICS) for interferon gamma (IFN-gamma) and/or interleukin (IL)-2 to HIV potential T-cell epitope (PTE) peptide pools representing Gag
Change in response rates of CD8 T-cell responses | Measured at Days 7, 14, 68, and 70
  Response rates of CD8 T-cell responses measured by ICS for IFN-gamma and/or IL-2 to HIV PTE peptide pools representing Gag
Change in response rates of T-cell responses | Measured at Days 7, 14, 68, and 70
  Response rates of T-cell responses as measured by IFN-gamma enzyme-linked immunospot (ELISpot) (at the option of the HVTN Laboratory Program)
Change in induction of binding antibodies to HIV-1 gag | Measured at Days 7, 14, and 70
  Induction of binding antibodies to HIV-1 gag

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fuchs, Study Chair — San Francisco Department of Public Health/University of California, San Francisco
Locations (4):
- United States (4):
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

REFERENCES:
- [Background] Rose NF, Marx PA, Luckay A, Nixon DF, Moretto WJ, Donahoe SM, Montefiori D, Roberts A, Buonocore L, Rose JK. An effective AIDS vaccine based on live attenuated vesicular stomatitis virus recombinants. Cell. 2001 Sep 7;106(5):539-49. doi: 10.1016/s0092-8674(01)00482-2. PMID 11551502
- [Background] Sacha JB, Chung C, Rakasz EG, Spencer SP, Jonas AK, Bean AT, Lee W, Burwitz BJ, Stephany JJ, Loffredo JT, Allison DB, Adnan S, Hoji A, Wilson NA, Friedrich TC, Lifson JD, Yang OO, Watkins DI. Gag-specific CD8+ T lymphocytes recognize infected cells before AIDS-virus integration and viral protein expression. J Immunol. 2007 Mar 1;178(5):2746-54. doi: 10.4049/jimmunol.178.5.2746. PMID 17312117
- [Background] Cooper D, Wright KJ, Calderon PC, Guo M, Nasar F, Johnson JE, Coleman JW, Lee M, Kotash C, Yurgelonis I, Natuk RJ, Hendry RM, Udem SA, Clarke DK. Attenuation of recombinant vesicular stomatitis virus-human immunodeficiency virus type 1 vaccine vectors by gene translocations and g gene truncation reduces neurovirulence and enhances immunogenicity in mice. J Virol. 2008 Jan;82(1):207-19. doi: 10.1128/JVI.01515-07. Epub 2007 Oct 17. PMID 17942549